CLINICAL TRIAL: NCT05271734
Title: Evaluation of the Compatibility of Different Eye Lid Retractors to the Direct Selective Laser Trabeculoplasty (DSLT) Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BelkinVision (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-02

CONDITIONS: OAG - Open-Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm -lid retractor placement (Experimental): Placement of a lid retractor the find out if the corneal limbus is exposed to 360 degrees
  Interventions: Device: Lid retractor placement

INTERVENTIONS:
Device: Lid retractor placement — Insertion of a lid retractor to find out if the corneal limbus is exposed in 360 degress

SUMMARY:
Direct Selective Laser Trabeculoplasty (DSLT) is an emerging therapeutic technology to treat glaucoma. DSLT was previously tested in 2 clinical trials and demonstrated promising safety and efficacy results in reducing the patient's intra ocular pressure.

Experience gained in the previous clinical studies indicates that a full exposure of the limbal area may be a challenge in patients with narrow palpebral fissures, narrow or floppy eyelids, and patients with deep-set eyes.

DETAILED DESCRIPTION:
The DSLT procedure is carried out in the doctor's office while the patient sits in front of the DSLT device (termed the "Eagle" device) for couple of minutes.

In this procedure, 120 laser applications are performed around the full circumference of the ocular limbus, after the system automatically recognizes the limbal target area. It is therefore essential that a full exposure of 3600 limbal area will be achieved, and this is done by placing an eye lid retractor (speculum) in the treated eye at the beginning of the procedure.

The purpose of this study is to evaluate the compatibility of different types of lid retractors. The lid retractors will be tested in adult volunteers visiting the study eye clinic for any reason.

ELIGIBILITY:
Inclusion Criteria.

* Adult volunteers (age ≥18 years old) of both sexes visiting the study eye clinic for any reason.
* Willing and able to participate in the study and to comply with the study procedures.
* Participant capable of giving informed consent.

Exclusion Criteria:

* Prior incisional ocular surgery or ocular trauma in the tested eye.
* Women who are pregnant.
* Any medical condition that interferes with the subject's ability to sit steady in front of the Eagle device.
* Known allergy to local anaesthesia eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Limbus Exposure | Baseline
  Full 360° Limbus exposure while subject is sitting.

CONTACTS AND LOCATIONS:
Locations (1):
- Akhali Mzera Eye Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No